CLINICAL TRIAL: NCT00396149
Title: A Phase I Study to Investigate the Safety, Tolerability and Pharmacodynamic Effects of SLIT(Tablets) With Recombinant Bet v1 Given in Single Rising Doses and in Higher Multi Dose Regimens to Subjects Sensitised to Birch Pollen
Brief Title: Safety, Tolerability and Pharmacodynamic Effects of Sublingual Immunotherapy (Tablets) With Recombinant Bet v1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Bruno ROBIN, Stallergenes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO49.06 DK
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2009-04

CONDITIONS: Birch Pollen-Related Rhinoconjunctivitis; Rhinitis, Allergic, Seasonal
Keywords: rBet v 1; Birch pollen allergy; Sublingual Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo group
  Interventions: Biological: Placebo
- Active group (Experimental): rBet v 1 tablets
  Interventions: Biological: rBet v 1

INTERVENTIONS:
Biological: Placebo — Two matching placebo tablets were administered every day over 2 weeks with a 2-day break for the week-end.
  Arms: Placebo
Biological: rBet v 1 — Two tablets (1 placebo + 1 rBet v 1 or 2 rBet v 1) were administered every day over 2 weeks with a 2-day break for the week-end. Administered doses ranged from 50 to 300 µg rBet v 1.
  Other Names: rBet v 1.0101
  Arms: Active group

SUMMARY:
To investigate the safety and tolerability of successive single rising doses of SLIT in subjects with allergic rhinitis and to investigate the safety and tolerability of multi high dose regimens of SLIT in subjects with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* Symptoms of birch pollen induced allergic rhinitis for at least the last 2 years.
* Sensitisation to birch pollen as demonstrated with a positive SPT to birch pollen and specific IgE level (birch pollen and r Bet v1) of at least Class 2 at screening.
* FEV1 at least of 80% of predicted values at screening.

Exclusion Criteria:

* Patient who previously received desensitization treatment to birch pollen and/or other betulaceae (e.g., hazel tree, alder…) or who plan to start desensitization treatment during this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Local tolerability | Assessed every day over 2 weeks
Global safety | Assessed every day over 2 weeks

SECONDARY OUTCOMES:
Immunological markers (IgE and IgG4) | Between selection and follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jorgen MALLING, Professor, Principal Investigator — National University Hospital, Copenhagen
Locations (1):
- National University Hospital - Allergy Unit 4222, Copenhagen, Denmark

REFERENCES:
- [Result] L. Winther, L.K. Poulsen, B. Robin, M. Mélac, H. Malling Safety and Tolerability of Recombinant Bet v 1 (rBet v 1) Tablets in Sublingual Immunotherapy (SLIT) The Journal of Allergy and Clinical Immunology February 2009 (Vol. 123, Issue 2, Page S215)